CLINICAL TRIAL: NCT03001492
Title: Does Measurement of Serum Progesterone on the Day of Trigger Matter?
Brief Title: Does Premature Luteinization Matter?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Osama Saber Thabet Abdalmageed, Lecturer of OBGYN, Women Health Hospital, Assiut Univerisity, Assiut University
Other Study IDs: Progesterone
Record Dates: First submitted 2016-12-17; First posted 2016-12-23 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Premature Progesterone Rise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Elevation of serum progesterone on the day of ovulation triggering in IVF/ICSI cycles is suggested to be associated with compromized outcomes. Others found that this rise didnot affect the IVF/ICSI outcomes. It is still controversal if premature luteinization would affect the IVF/ICSI outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Planned fresh Embryo transfer

Exclusion Criteria:

* Cancelation of the embryo transfer for any reason

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All the women undergo controlled ovarian hyperstimulation for IVF/ICSI. only fresh cycles will be involved
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnacy rate | 14 days after the day of embryo transfer (ET)

CONTACTS AND LOCATIONS:
Overall Officials: Osama Abdalmageed, Principal Investigator — Women health center
Locations (1):
- Osama Abdalmageed, Asyut, Non-US/Non-Canadian, Egypt

REFERENCES:
- [Background] Sonmezer M, Pelin Cil A, Atabekoglu C, Ozkavukcu S, Ozmen B. Does premature luteinization or early surge of LH impair cycle outcome? Report of two successful outcomes. J Assist Reprod Genet. 2009 Mar;26(2-3):159-63. doi: 10.1007/s10815-009-9299-5. Epub 2009 Feb 18. PMID 19224360